CLINICAL TRIAL: NCT06996782
Title: A Phase Ib/II Open-Label, Multicentre Platform Study Evaluating Novel Combinations in Participants With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Platform Study in Non-Small Cell Lung Cancer (NSCLC)
Acronym: ALTAIR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D702KC00001; 2024-519786-22 (Other: EU CT number)
Record Dates: First submitted 2025-05-05; First posted 2025-05-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: Checkpoint inhibitor (CPI); Platinum-based chemotherapy; T-cell immunoreceptor with lg and Immunoreceptor Tyrosine-based Inhibition Motif (ITIM) domains (TIGIT); Programmed death-ligand 1 (PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub study 2 Part A: Safety run-in (Experimental): Participants with squamous and non-squamous NSCLC will receive combination therapy of rilvegostomig, ramucirumab, and platinum-based chemotherapy to assess the safety and tolerability of this regimen.
  Interventions: Drug: Rilvegostomig; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Ramucirumab
- Sub study 2 Part B: Dose expansion (Experimental): Participants will be randomised 1:1 into one of 2 treatment arms (rilvegostomig + chemotherapy + ramucirumab OR rilvegostomig + chemotherapy) in non-squamous histology cohorts and into a single arm (rilvegostomig + chemotherapy+ ramucirumab) in squamous histology cohorts.
  Interventions: Drug: Rilvegostomig; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Ramucirumab

INTERVENTIONS:
Drug: Rilvegostomig — Rilvegostomig will be administered as an intravenous (IV) infusion.
  Other Names: AZD2936
Drug: Cisplatin — Cisplatin will be administered as SoC as an IV infusion.
Drug: Carboplatin — Carboplatin will be administered as SoC as an IV infusion.
Drug: Pemetrexed — Pemetrexed will be administered as SoC as an IV infusion.
Drug: Paclitaxel — Paclitaxel will be administered as SoC as an IV infusion.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered as SoC as an IV infusion.
Drug: Ramucirumab — Ramucirumab will be administered as an IV infusion.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of multiple study interventions including novel-novel combinations or novel agents in combination with standard therapy for the treatment of metastatic NSCLC.

DETAILED DESCRIPTION:
This is a multicentre, open-label study to evaluate the safety and efficacy of various combinations of study interventions in participants with advanced or metastatic NSCLC (mNSCLC).

The study will include a sub-study (sub-study 2) focused on a specific treatment that may include 2 parts -

1. Part A consisting of one of more safety run-in cohorts to evaluate 2 or more dose levels to identify the recommended Phase 2 dose (RP2D) unless RP2D has been established then Part A will not be required; and
2. Part B consisting of one or more expansion cohorts.

The originally planned Sub-study 1 was withdrawn (cancelled) and will not be conducted.

Sub-study 2 will evaluate the safety, tolerability, and anti-tumour activity of rilvegostomig plus standard of care (SoC) platinum-based chemotherapy, with or without ramucirumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed squamous or non-squamous NSCLC with a current Stage IV mNSCLC.
* Provision of acceptable archival tumour tissue (or fresh tumour tissue biopsy if archival tumour tissue is not available and if clinically feasible) is mandatory at screening.
* Measurable disease as defined by at least one lesion that can be accurately measured at baseline as ≥ 10 mm at the longest diameter.
* Minimum life expectancy of 12 weeks in the opinion of the investigator.
* Adequate organ and marrow function.
* Contraceptive use by male or female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Adequate organ and marrow function.

Inclusion Criteria for Sub Study 2:

* Programmed death-ligand 1 (PD-L1) tumour proportion score (TPS) ≥ 1% (per local report).
* Adequate coagulation and urinalysis.
* Minimum body weight of 30 kg.

Exclusion Criteria:

* Participants with epidermal growth factor receptor mutations, anaplastic lymphoma receptor fusions or any other known genomic alteration for which targeted therapy is approved in the first line per local standard of care.
* Presence of small cell and neuroendocrine histology components.
* Any severe or uncontrolled systemic diseases, including uncontrolled hypertension, and active bleeding diseases, ongoing or active known infection; interstitial lung disease/pneumonitis (of any grade); unstable and/or symptomatic venous thromboembolism, serious chronic gastrointestinal conditions associated with diarrhoea, active non-infectious skin disease or substance abuse.
* Has had a prior stem cell, bone marrow, allogenic tissue, or solid organ transplant.
* Has an active autoimmune disease that has required systemic treatment in the past 5 years.
* History of clinically significant arrhythmia, cardiomyopathy of any aetiology or symptomatic congestive heart failure.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention or presence of small cell and neuroendocrine histology components.
* Persistent toxicities (common terminology criteria for adverse events [CTCAE] ≥ Grade 2) caused by previous anti-cancer therapy, excluding alopecia.
* Spinal cord compression or symptomatic brain metastases.
* Treatment with any other anti-cancer agents or immunosuppressive medication.
* Palliative radiotherapy with a limited field of radiation within 2 weeks or with a wide field of radiation or to more than 30% of the bone marrow within 4 weeks, prior to the first dose of study intervention.

Exclusion Criteria for Sub Study 2:

* Known active hepatitis A.
* Acute hepatitis B infection (anti-hepatitis B core antibody [HBc] immunoglobulin M [IgM] positive) or chronic hepatitis B infection with HBV DNA ≥ 2000 IU/mL.
* Active hepatitis C infection (anti-HCV positive with HCV RNA detectable) or anti- HCV positive with HCV RNA undetectable for less than 12 weeks following treatment for HCV.
* Known human immunodeficiency virus (HIV) infection that is not well controlled.
* Evidence of Grade ≥ 1 central nervous system (CNS) haemorrhage.
* Uncontrolled arterial hypertension ≥ 150 mm Hg (systolic) and/or ≥ 100 mm Hg (diastolic).
* Has radiologically documented evidence of major blood vessel invasion or encasement by cancer, or major airway invasion by cancer or intra-tumour cavitation.
* Has experienced any arterial thrombotic event, a Grade ≥ 3 bleeding event or has gross haemoptysis.
* Has significant bleeding disorders, serious or nonhealing wound, ulcer or clinically relevant congestive heart failure.
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection.
* Has cirrhosis at a level of Child-Pugh B (or worse), or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
* Prior systemic therapy received for advanced or mNSCLC.
* Prior exposure to an anti-T-cell immunoreceptor with Ig and Immunoreceptor Tyrosine-based Inhibition Motif domains (TIGIT) therapy or immune-oncology agent such as anti-programmed cell death protein 1 (PD-1), anti-PD-L1, or anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4), or any other anti-cancer therapy targeting immune-regulatory receptors or mechanisms.
* Chronic therapy with antiplatelet agents.
* Prior exposure to anti-vascular endothelial growth factor (VEGF) therapy.
* Medical contraindication to protocol-specified platinum doublet regimens or ramucirumab.
* Known allergy or hypersensitivity to rilvegostomig or any of the excipients of rilvegostomig, cisplatin, carboplatin, paclitaxel or nab-paclitaxel or pemetrexed or ramucirumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-02-23 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Approximately 46 months
  To assess the safety and tolerability and determine RP2D of the combination of novel anti-cancer agents.
Part A: Number of partcipants with dose limiting toxicity (DLT) | Approximately 46 months
  To assess the safety and tolerability and determine RP2D of the combination of novel anti-cancer agents.
Part B: Objective response (OR) | Approximately 46 months
  The OR is defined as a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR).

SECONDARY OUTCOMES:
Part A: Objective response (OR) | Approximately 46 months
  The OR is defined as a BOR of confirmed CR or confirmed PR.
Part A and Part B: Duration of response (DOR) | Approximately 46 months
  The DoR is defined as the time from the date of first documented objective response (which is subsequently confirmed) until date of first documented disease progression or death (by any cause in the absence of disease progression).
Part A and Part B: Time to response (TTR) | Approximately 46 months
  Time to response is defined as the time from the start of treatment until the date of first documented response.
Part A and Part B: Disease control (DC) | Approximately 46 months
  Disease control is defined as if a participant has a best overall response of confirmed CR or confirmed PR or who have stable disease (SD) for at least 7 weeks after start of treatment.
Part A and Part B: Progression free survival (PFS) | Approximately 46 months
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from assigned therapy or receives another anti-cancer therapy prior to progression.
Part A and Part B: Progression free survival at 6 months (PFS6) | From Day 1 pre-dose to 6 months
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from assigned therapy or receives another anti-cancer therapy prior to progression.
Part A and Part B: Progression free survival at 12 months (PFS12) | From Day 1 pre-dose to 12 months
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from assigned therapy or receives another anti-cancer therapy prior to progression.
Part A and Part B: Overall survival (OS) | Approximately 46 months
  Overall survival is defined as the time from the start of treatment until death due to any cause regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy.
Part A and Part B: Overall survival at 12 months (OS12) | From Day 1 pre-dose to 12 months
  Overall survival is defined as the time from the start of treatment until death due to any cause regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy.
Part A and Part B: Serum concentration | Approximately 46 months
  To assess the serum concentration of the novel anti-cancer agents in combination.
Part A and Part B: Maximum plasma drug concentration (Cmax) | Approximately 46 months
  To assess the Cmax of the novel anti-cancer agents in combination.
Part A and Part B: Area under plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) | Approximately 46 months
  To assess the AUClast of the novel anti-cancer agents in combination.
Part A and Part B: Area under plasma concentration-time curve from time 0 to infinity (AUC∞) | Approximately 46 months
  To assess the AUC∞ of the novel anti-cancer agents in combination.
Part A and Part B: Time to reach maximum concentration following drug administration (tmax) | Approximately 46 months
  To assess the tmax of the novel anti-cancer agents in combination.
Part A and Part B: Terminal elimination half-life (t1/2λz) | Approximately 46 months
  To assess the t1/2λz of the novel anti-cancer agents in combination.
Part A and Part B: Clearance (CL) | Approximately 46 months
  To assess the CL of the novel anti-cancer agents in combination.
Part A and Part B: Volume of distribution at terminal phase (Vz) | Approximately 46 months
  To assess the Vz of the novel anti-cancer agents in combination.
Part A and Part B: Number of participants with anti-drug antibodies (ADAs) | Approximately 46 months
  To assess the immunogenicity of the novel anti-cancer agents in combination.

CONTACTS AND LOCATIONS:
Locations (86):
- United States (9):
  - Research Site, Phoenix, Arizona
  - Research Site, Santa Rosa, California
  - Research Site, Jacksonville, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Cleveland, Ohio
  - Research Site, Providence, Rhode Island
  - Research Site, Tyler, Texas
- Belgium (3):
  - Research Site, Anderlecht
  - Research Site, Hasselt
  - Research Site, Leuven
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Fortaleza
  - Research Site, Natal
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- China (10):
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Deyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Wuhan
- France (7):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (5):
  - Research Site, München
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Würzburg
- Italy (4):
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Pavia
  - Research Site, Roma
- Japan (7):
  - Research Site, Bunkyō City
  - Research Site, Kashiwa
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Niigata
  - Research Site, Shinjuku-ku
  - Research Site, Toyoake-shi
- Malaysia (4):
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
  - Research Site, Singapore
- Research Site, Chisinau, Moldova
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Leiden
- Research Site, Lima, Peru
- Poland (3):
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Olsztyn
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
- South Korea (2):
  - Research Site, Seongbuk-Gu
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Rachathewi
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Fatih
  - Research Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/